CLINICAL TRIAL: NCT03474029
Title: Six Weeks of Daily Rifapentine vs. a Comparator Arm of 12-16 Week Rifamycin-based Treatment of Latent M. Tuberculosis Infection: Assessment of Safety, Tolerability and Effectiveness
Brief Title: Assessment of the Safety, Tolerability, and Effectiveness of Rifapentine Given Daily for LTBI
Acronym: ASTERoiD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-7024
Record Dates: First submitted 2018-03-08; First posted 2018-03-22 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Latent Tuberculosis
Keywords: latent tuberculosis; rifapentine
MeSH Terms: conditions — Latent Tuberculosis | interventions — rifapentine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 6 weeks of daily rifapentine (6wP) (Experimental): Rifapentine daily for 6 weeks: 600 mg of Rifapentine (RPT) given once daily for 6 weeks
  Interventions: Drug: Rifapentine daily for 6 weeks
- 12-16 week rifamycin-based regimen (Active Comparator): A 12-16 week rifamycin-based regimen available at the participant's site:
  "Rifapentine and Isoniazid weekly for 12 weeks" (3HP) or "Rifampin and Isoniazid daily for 12 weeks" (3HR) or "Rifampin daily for 16 weeks" (4R)
  Interventions: Drug: Rifapentine and Isoniazid weekly for 12 weeks; Drug: Rifampin and Isoniazid daily for 12 weeks; Drug: Rifampin daily for 16 weeks

INTERVENTIONS:
Drug: Rifapentine daily for 6 weeks — 600 mg of Rifapentine (RPT) given once daily (o.d., omni die) for 6 weeks (6wP).
  Other Names: priftin
  Arms: 6 weeks of daily rifapentine (6wP)
Drug: Rifapentine and Isoniazid weekly for 12 weeks — Rifapentine (RPT) 900 mg and isoniazid (INH) 900 mg given once-weekly for 12 weeks (3HP).*
  *Dose adjustments based on patient's weight will be made according to ATS/CDC/IDSA guidelines.
  RPT 900 mg once-weekly for persons weighing > 50 kg. For persons weighing < 50 kg, the following doses will be given: weight > 25-32 kg - RPT 600 mg; weight > 32-50 kg - RPT 750 mg; + INH 15 mg/kg (round up to nearest 50 or 100 mg; 900 mg max).
  Arms: 12-16 week rifamycin-based regimen
Drug: Rifampin and Isoniazid daily for 12 weeks — Rifampin (RIF) 600 mg and Isoniazid (INH) 300 mg given once-daily for 12 weeks (3HR)*.
  *Dose adjustments based on patient's weight will be made according to ATS/CDC/IDSA guidelines.
  RIF 600 mg daily for persons weighing > 50 kg. For persons weighing < 50 kg, give 10 mg/kg daily; round up to nearest 50 or 100 mg; + INH 5 mg/kg daily (rounded up to nearest 50 or 100 mg; 300 mg max).
  Arms: 12-16 week rifamycin-based regimen
Drug: Rifampin daily for 16 weeks — Rifampin (RIF) 600 mg given once-daily for 16 weeks (4R).*
  *Dose adjustments based on patient's weight will be made according to ATS/CDC/IDSA guidelines.
  RIF 600 mg daily for persons weighing > 50 kg. For persons weighing < 50 kg, 10 mg/kg daily; round up to nearest 50 or 100 mg.
  Arms: 12-16 week rifamycin-based regimen

SUMMARY:
This study is conducted to compare the safety and effectiveness of a novel short 6-week regimen of daily rifapentine (6wP, experimental arm) with a comparator arm of 12-16 weeks of rifamycin-based treatment (standard of care, control arm) of latent M. tuberculosis infection (LTBI).

This trial is conducted among persons who are at increased risk of progression to tuberculosis (TB) and require treatment of LTBI. The study will be conducted in low, medium and high TB incidence settings that have treatment of LTBI as their standard of care and offer 12-16 week rifamycin-based therapy as standard of care.

The hypothesis of this study is that the safety and effectiveness of the experimental treatment (6wP arm) is non-inferior to a comparator arm of 12-16 weeks of rifamycin-based treatment of LTBI (control arm).

Participants are enrolled and randomly assigned to one of the two study arms: experimental 6wP or control. The comparator (control) arm's treatment regimens include 12 weeks of once-weekly isoniazid (INH) and rifapentine (3HP), 12 weeks of daily INH and rifampin (3HR), and 16 weeks of daily rifampin (4R). A total of 560 participants per arm (1,120 total) for the evaluation of safety and 1,700 participants per arm (3,400 total) for the evaluation of effectiveness will be enrolled, given treatment as per randomization assignment, and followed for 24 months from the date of enrollment.

After completion of data collection, statistical analyses will be conducted to compare proportions of drug discontinuation due to adverse drug reaction (ADR) and proportions of newly diagnosed tuberculosis between 6wP and control arm.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females > 12 years old. Women of child-bearing potential who are not surgically sterilized must agree to practice an adequate method of contraception (barrier method or non-hormonal intrauterine device) or abstain from heterosexual intercourse during study drug treatment.
* Persons with LTBI who do not have evidence of TB disease and are at increased risk of progression to TB. M. tuberculosis infection may be demonstrated by either a positive tuberculin skin test (TST) or a positive interferon gamma release assay (IGRA; e.g., QuantiFERON or T.SPOT.TB). Persons with LTBI at increased risk of progression to TB are those with one of the following:

  1. Household and other close contacts (> 4 hours of exposure in a one week period) within 2 years prior to enrollment, of persons with culture-confirmed TB A positive nucleic acid amplification test (NAAT)/GeneXpert in the source case may be used for enrollment prior to culture confirmation
  2. Recent M. tuberculosis infection, defined as converting from a documented negative to positive TST or IGRA within 2 years prior to enrollment. Persons without known close contact to someone with active pulmonary TB who have a conversion by IGRA may require additional evaluation to rule out a false conversion.
  3. HIV co-infection (with CD4+ T-lymphocyte count > 100 cells/mm3).
  4. ≥ 2 cm2 of pulmonary parenchymal fibrosis on chest X-ray and no prior history of treatment for TB or LTBI.
  5. Recent (within 3 years prior to enrollment) immigration to the United States or other country with low to moderate TB incidence, with abnormal chest X-ray, and no evidence of active TB.
  6. Recent (within 2 years prior to enrollment) immigration to the United States or other country with low to moderate TB incidence, from a country with an estimated incidence rate of TB > 150 per 100,000
  7. An increased risk of TB due to medical conditions such as end-stage renal disease, or due to use of immunosuppressive medications such as chronic steroids or TNF-alpha inhibitors.
* Willing to provide signed informed consent, or parental permission and participant assent.

Exclusion Criteria:

* Current confirmed culture-positive or clinical TB.
* Suspected current TB. Includes cases in which active TB cannot be eliminated as a possibility (by the site investigator)
* TB resistant to any rifamycin in the source case
* A history of treatment for > 7 consecutive days with a rifamycin or > 30 consecutive days with INH within 2 years prior to enrollment.
* A documented history of completing an adequate course of treatment for TB disease or LTBI in a person who is HIV-seronegative.
* History of allergy or intolerance to rifamycins.
* Serum alanine aminotransferase (ALT; SGPT) or serum aspartate aminotransferase (AST; SGOT) > 5x upper limit of normal among persons in whom baseline ALT or AST is determined+.
* HIV-seropositive and on antiretroviral therapy that cannot be given with rifampin or rifapentine due to drug-drug interactions.
* Receiving concomitant medications that are known to be contraindicated with any study drug.
* Females who are currently pregnant, breastfeeding, or intend to become pregnant within 120 days of enrollment.
* Weight < 25 kg.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Treatment discontinuation due to adverse drug reaction | from the date of enrollment to the date of scheduled completion of assigned treatment
  Safety outcome. Drug discontinuation due to adverse drug reaction (ADR) associated with experimental treatment (6wP) or active comparator treatment (the rifamycin-based 3HP, 3HR, or 4R). Attribution of an adverse event (AE) to study drugs will be initially determined by the local site investigator, reviewed by an independent, blinded adjudication panel and with final attribution determined by the sponsor.
Culture-confirmed tuberculosis (TB) in participants 18 years old and older and culture-confirmed or clinical TB in participants less then 18 years old. | within 24 months from the date of enrollment
  Effectiveness outcome. Culture-confirmed tuberculosis (TB) in participants 18 years old and older and culture-confirmed or clinical TB in participants less then 18 years old. Diagnosis of culture-confirmed TB will be performed using liquid and/or solid media methods.

SECONDARY OUTCOMES:
Proportion who complete assigned treatment | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
Proportion with drug discontinuation for any reason | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
Proportion with any grade 3, 4, or 5 (i.e., death) adverse event associated with study drug | within 6 months from the date of enrollment
Proportion who have died for any reason | within 24 months from the date of enrollment
Proportion with hepatitis and non-hepatotoxic systemic drug reactions | within 6 months from the date of enrollment
Proportion with culture-confirmed or clinical TB regardless of age | within 24 months from the date of enrollment
Proportion with TB among those who complete assigned therapy | within 24 months from the date of enrollment
Safety (defined as treatment discontinuation due to adverse drug reaction) among participants with human immunodeficiency virus (HIV) infection. | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
  Proportion of HIV-infected patients with drug discontinuation due to adverse drug reaction (ADR) associated with experimental treatment (6wP) or active comparator treatment (the rifamycin-based 3HP, 3HR, or 4R) . Attribution of an adverse event (AE) to study drugs will be determined by the local site investigator.
Safety (defined as treatment discontinuation due to adverse drug reaction) among participants < 18 years old. | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
  Proportion of participants < 18 years old with drug discontinuation due to adverse drug reaction (ADR) associated with experimental treatment (6wP) or active comparator treatment (the rifamycin-based 3HP, 3HR, or 4R) . Attribution of an adverse event (AE) to study drugs will be determined by the local site investigator.
Tolerability (defined as proportion of with drug discontinuation for any reason) among participants with human immunodeficiency virus (HIV) infection. | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
  Proportion of HIV-infected patients with drug discontinuation for any reason
Tolerability (defined as proportion of with drug discontinuation for any reason) among participants < 18 years old. | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
  Proportion of participants < 18 years old with drug discontinuation for any reason
Effectiveness among participants with human immunodeficiency virus (HIV) infection. | within 24 months from the date of enrollment
  Proportion of HIV-infected patients with culture-confirmed tuberculosis (TB) in participants 18 years old and older and culture-confirmed or clinical TB in participants less then 18 years old. Diagnosis of culture-confirmed TB will be performed using liquid and/or solid media methods.
Effectiveness among participants < 18 years old. | within 24 months from the date of enrollment
  Proportion of participants < 18 years old with culture-confirmed tuberculosis or clinical TB. Diagnosis of culture-confirmed TB will be performed using liquid and/or solid media methods.

OTHER OUTCOMES:
Proportions of drug discontinuation due to adverse drug reactions in experimental (6wP) arm and each treatment regimen in the comparator arm: 3HP, 3HR, 4R | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
Proportions of treatment discontinuations for any reason in experimental (6wP) arm and each treatment regimen in the comparator arm: 3HP, 3HR, 4R | from date of enrollment until the maximum accepted time for treatment completion as follows: 9 weeks for 6wP treatment, 16 weeks for 3HP, 16 weeks for 3HP, and 21 weeks for 4R
Effectiveness of experimental (6wP) arm and each treatment regimen in the comparator arm: 3HP, 3HR, 4R | within 24 months from the date of enrollment
  Proportion of participants with culture-confirmed tuberculosis (TB) in participants 18 years old and older and culture-confirmed or clinical TB in participants less then 18 years old. Diagnosis of culture-confirmed TB will be performed using liquid and/or solid media methods.
Proportion with resistance to rifamycins or isoniazid among persons who develop TB to each regimen in the comparator arm: 3HP, 3HR, 4R. | within 24 months from the date of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Sterling, MD, Study Chair — Vanderbilt University Medical Center, USA; Robert Belknap, MD, Study Chair — Denver Public Health (USA); Amber Robinson, PhD, Study Director — Centers for Disease Control and Prevention; Rosanna M Boyd, PhD, Study Director — Centers for Disease Control (USA); Dick Menzies, MD, Study Chair — McGill University
Locations (16):
- United States (7):
  - Denver Health and Hospital Authority, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - New York Harbor Healthcare System, Manhattan, New York
  - New York City Bureau of TB Control, New York, New York
  - San Antonio VA, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Australia (3):
  - Liverpool Hospital, Sydney
  - Paramatta Chest, Sydney
  - Royal Prince Alfred Hospital, Sydney
- Canada (5):
  - Calgary TB Clinic, Calgary, Alberta
  - Edmonton TB Clinic, Edmonton, Alberta
  - British Columbia Centre for Disease Control, Vancouver, British Columbia
  - Toronto Western Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Desmond Tutu TB Center, Stellenbosch, South Africa

REFERENCES:
- See also: Tuberculosis Trials Consortium (TBTC) — https://www.cdc.gov/tb/research/tbtc.html